CLINICAL TRIAL: NCT06015126
Title: Efficacy and Safety of Metronomic Oral Vinorelbine Plus Anlotinib in HER2-negative Metastatic Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yan Xue (Other)
Responsible Party: Sponsor-Investigator, Yan Xue, Director of tumor hospital, Xi'an International Medical Center Hospital
Organization: Xi'an International Medical Center Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y-pierrefabre202102-0108
Record Dates: First submitted 2023-08-08; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Label 1 (Experimental): metronomic oral vinorelbine plus anlotinib
  Interventions: Drug: metronomic oral vinorelbine plus anlotinib

INTERVENTIONS:
Drug: metronomic oral vinorelbine plus anlotinib — To clarify the efficacy and safety of metronomic oral vinorelbine plus anlotinib in HER2-negative metastatic breast cancer patients, adding new data for the posterior treatment of HER2-negative advanced breast cancer

SUMMARY:
vinorelbine are one of the main chemotherapy drugs used in the treatment of advanced breast cancer. It is available in oral form, making it convenient to use and an ideal choice for rhythmic chemotherapy. In advanced breast cancer,metronomic oral vinorelbine chemotherapy has been the subject of several clinical studies, with proven effectiveness and good safety, showing great prospects for application.

Considering the current lack of targeted, efficient, and convenient drugs for HER2-negative advanced breast cancer in later lines of treatment, and based on the preliminary efficacy of metronomic oral vinorelbine, anlotinib, and rhythmic chemotherapy in breast cancer, we plan to explore the efficacy and safety of combining metronomic oral vinorelbine chemotherapy with anlotinib in the treatment of HER2-negative advanced breast cancer, providing new data for the treatment of HER2-negative advanced breast cancer.

DETAILED DESCRIPTION:
Research Title A single-center, open-label, single-arm clinical study on the efficacy and safety of Changchun Ruibin rhythmic chemotherapy combined with anlotinib in HER2-negative advanced breast cancer.

Study Drugs - metronomic oral vinorelbine: 30mg/capsule, 20mg/capsule - Anlotinib: 12mg/capsule, 10mg/capsule, 8mg/capsule

Research Objective To determine the efficacy and safety of metronomic oral vinorelbine chemotherapy combined with anlotinib in the treatment of HER2-negative advanced breast cancer, and to provide new data for later-line treatment of HER2-negative advanced breast cancer.

Study Design A single-center, open-label, single-arm clinical study with a planned enrollment of 60 patients.

ELIGIBILITY:
Inclusion Criteria：

* Voluntarily sign an informed consent form;
* Females aged 18 years or older;
* ECOG physical performance status score of 0-2;
* Histologically confirmed HER2-negative metastatic breast cancer patients, and patients with locally recurrent disease who cannot undergo curative surgery or radiation therapy;
* HR-positive/HER2-negative advanced breast cancer patients who have primary endocrine resistance or disease progression after first-line endocrine ± targeted therapy;
* Triple-negative advanced breast cancer patients with disease progression after first-line chemotherapy ± immunotherapy;
* Blood routine examination meets the following conditions: ①absolute neutrophil count (ANC) ≥1.5×10^9/L, ② platelets ≥100×10^9/L, ③ hemoglobin ≥90 g/L, ④ white blood cell count ≥3.0×10^9/L;
* The liver function meets the following criteria: ① serum total bilirubin ≤ 1.5 × ULN, and if there is liver metastasis, it should be ≤ 3 × ULN; ② AST or ALT ≤ 3 × ULN, and if there is liver metastasis, it should be ≤ 5 × ULN;
* The renal function meets the following criteria: serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min (calculated according to the Cockroft-Gault formula);
* Female patients who meet the following criteria can participate in this study: ① Patients are not capable of reproduction; ② Patients have reproductive capacity, and have a negative result on the pregnancy test within 7 days before the first administration of the investigational drug, are not in the lactation period, and continuously adopt effective contraceptive measures before entering the study and during the entire study period and within 6 months after the last administration of the investigational drug.

Exclusion Criteria:

* Patients who have previously received treatment with vinorelbine and/or anlotinib;
* Patients with active or untreated brain metastasis;
* Patients who have had or currently have other malignancies within 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invades basement membrane)];
* Patients who have undergone major surgery (including thoracotomy biopsy) or suffered a significant trauma (such as bone fracture) within 4 weeks before randomization, have unhealed wounds or fractures at the time of screening, or are expected to undergo major surgery during the study period;
* Patients with a history of myocardial infarction within the past 6 months; history of congestive heart failure with New York Heart Association (NYHA) classification ≥ II, or severe arrhythmia (excluding atrial fibrillation and paroxysmal supraventricular tachycardia) that cannot be controlled by medication;
* Patients with known allergies to the drugs and their excipients involved in this trial;
* Patients with a known history of hypersensitivity reactions to any investigational drugs;
* Patients who are simultaneously participating in other trials;
* Patients who cannot evaluate the efficacy of the treatment plan with existing technology;
* Patients judged unsuitable for participation by other investigators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  It is an indicator of the long-term efficacy of the drug.

SECONDARY OUTCOMES:
Objective Response Rate | 4 weeks
  The proportion of patients with the best response of complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST).
Disease Control Rate | 4 weeks
  The proportion of patients with tumor shrinkage or stability maintained for a certain period, including cases of CR, PR, and stable disease (SD).
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  It is an indicator of the long-term efficacy of the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Xue, Principal Investigator — Xi'an International Medical Center Hospital
Locations (1):
- Xi'an International Medical Center Hospital, Xi'an, Shaanxi, China